CLINICAL TRIAL: NCT02462954
Title: A Phase I Safety Study Of The Caya® Diaphragm Used With ContraGel®
Brief Title: A Safety Study Of The Caya® Diaphragm Used With ContraGel®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A13-127
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Contraception
Keywords: Contraception; Vaginal Gel; Diaphragm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ContraGel (Experimental): ContraGel, a personal lubricant has a Conformite Europeenne (CE) mark and has been used with barrier devices in Europe and other countries outside the US, but it is not currently approved by the US FDA.
  Interventions: Device: ContraGel
- HEC Placebo (Placebo Comparator): The placebo gel is supplied by CONRAD in pre-filled individual applicators, each applicator containing 4.0 mL of HEC gel. Placebo gel contains HEC as the gel thickener, purified water, sodium chloride, sorbic acid and sodium hydroxide.
  Interventions: Device: HEC Universal Placebo gel

INTERVENTIONS:
Device: ContraGel
  Arms: ContraGel
Device: HEC Universal Placebo gel
  Arms: HEC Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of ContraGel versus the hydroxyethylcellulose (HEC) Universal Placebo gel when used with the Caya diaphragm during two 7-day periods of daily use, the first without intercourse and the second with intercourse.

DETAILED DESCRIPTION:
This single-center randomized, parallel, Phase I study will compare the safety of ContraGel delivered by the Caya diaphragm versus HEC universal placebo gel delivered by the Caya diaphragm in approximately 24 healthy premenopausal women protected from pregnancy by female sterilization. Women will use the assigned product during two 7-day periods of daily use, the first without intercourse and the second with intercourse.

Each woman will be seen in approximately 6 visits and will be contacted via one scheduled follow-up call after Visit 6.

At Visit 1, volunteers will be consented and undergo procedures to confirm they are eligible to continue in the study.

At Visit 2, once it has been confirmed that the participant meets all of the inclusion criteria and none of the exclusion criteria, baseline genital tract samples will be taken.

At Visit 3,baseline genital tract samples will be taken for Test Cycle 1 (before product use with no intercourse). Participants will be randomized in a 1:1 ratio to insert the Caya diaphragm to deliver either ContraGel or the HEC placebo every day for two 7-day periods in two separate menstrual cycles. The participant will receive study supplies. She will be instructed to refrain from intercourse during the first 7-day period and to insert the Caya each day for between 6-12 hours. She will be instructed to return to the clinic at Visit 4 with the diaphragm in place.

At Visit 4, genital tract samples will be taken after 7 days of product use without intercourse (Test Cycle 1).

At Visit 5, baseline genital tract samples will be taken for Test Cycle 2 (before product use with intercourse). The participant will receive study supplies and will be instructed to engage in two sex acts during this 7-day period, the second sex act to take place using the study products 6-12 hours prior to Visit 6. Participants will be instructed to return to the clinic at Visit 6 with the diaphragm still in place.

At Visit 6, genital tract samples will be taken after 7 days of product use with intercourse (Test Cycle 2).

A follow-up call/contact will be scheduled for 1 to 2 weeks after Visit 6. The participant will be asked about any adverse events (AEs) experienced and medications taken since the last visit. The participant will then be exited from the study, unless she has symptoms that require follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet all of the following criteria prior to genital sampling at Visit 2.

  * Age 18-50 years, inclusive
  * General good health, by volunteer history and per investigator judgment
  * History of regular menstrual cycles of 24-35 days (inclusive), by volunteer report
  * History of Pap smears and follow-up consistent with standard medical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1.
  * Willing to abstain from and engage in intercourse and abstain from the use of vaginal products as required in the protocol
  * In a mutually monogamous relationship for at least the last four months with a male partner who:

    * Is at least 18 years old
    * Is willing and able to comply with protocol requirements including sexual activity/abstinence requirements
    * Can engage in vaginal intercourse with the participant without condoms, as specified in protocol
    * Has no known risk for sexually transmitted infections (STIs)
    * Has no known history of sensitivity/allergy to any component of ContraGel, HEC placebo gel, silicone or nylon
  * Protected from pregnancy by female sterilization
  * Vaginal and cervical anatomy that, in the opinion of the investigator, lends itself to easy colposcopy and genital tract sample collection
  * Willing to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* Volunteers must meet none of the following criteria prior to genital sampling at Visit 2.

  * History of hysterectomy
  * Currently pregnant or within two calendar months from the last pregnancy outcome. Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome.
  * Current use of any hormonal contraceptive (oral, transdermal, transvaginal, implant, or hormonal intrauterine contraceptive device) or a copper intrauterine device (IUD), or use of Depo-Provera in the last 6 months
  * Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
  * Significant gynecological abnormalities (including abnormal vaginal bleeding or excessive vaginal discharge)
  * Caya diaphragm does not appropriately fit volunteer, as determined by clinician
  * Inability to insert, position, and/or remove Caya diaphragm by volunteer
  * History of sensitivity/allergy to any component of ContraGel, HEC placebo gel, K-Y® Jelly, topical anesthetic, silicone or nylon, and to both silver nitrate and Monsel's solution
  * In the last six months, either the volunteer or her male partner diagnosed with or treated for any STI or pelvic inflammatory disease by self report. Note: Women with a history of genital herpes or condylomata who have been asymptomatic for at least six months may be considered for eligibility
  * Nugent score greater than or equal to 7
  * Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, or HIV
  * Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for a sexually transmitted infection
  * Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
  * Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
  * Known current drug or alcohol abuse which could impact study compliance
  * Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
  * History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
  * Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, or antivirals (e.g. acyclovir or valacyclovir). Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use Tylenol on an as-needed but not daily basis during the study
  * Grade 2 or higher abnormality per the November 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading of the Severity of Adverse Events or clinically significant lab abnormalities as determined by clinician
  * Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or her male partner which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse experiences (TEAEs) among female participants: urogenital, product-related, and/or serious | after two 7-day periods of daily use, the first without intercourse and the second with intercourse
Changes from baseline in the following safety endpoints [composite]: | after two 7-day periods of daily use, the first without intercourse and the second with intercourse
  * Findings on pelvic exam, including colposcopy
  * Vaginal pH (measure of acidity and alkalinity), Nugent score, and microflora
  * Anti-bacterial activity in cervicovaginal fluid (CVF)
  * Soluble markers of inflammation in cervicovaginal fluid (CVF)
  * Epithelial integrity and immune cell activation/phenotype in genital tissues
  * Findings on pelvic exam, including colposcopy
  * Vaginal pH, Nugent score, and microflora
  * Anti-bacterial activity in cervicovaginal fluid (CVF)
  * Soluble markers of inflammation in cervicovaginal fluid (CVF)
  * Epithelial integrity and immune cell activation/phenotype in genital tissues

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mauck, Study Director — CONRAD
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurman A, Cunningham T, Fichorova R, Herold BC, Hillier SL, Chandra N, Doncel GF. A phase I randomized safety study of a single-size silicone rubber diaphragm used with or without a lactic-acid-containing diaphragm gel. Contraception. 2019 Dec;100(6):430-437. doi: 10.1016/j.contraception.2019.06.004. Epub 2019 Aug 21. PMID 31442441